CLINICAL TRIAL: NCT04772469
Title: Self-Test Strategies and Linkage Incentives to Improve ART and PrEP Uptake in Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Pennsylvania (Other); Impact Research & Development Organization (Other); National Institute of Mental Health (NIMH) (NIH); Duke University (Other); Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-28205; 1R01MH120176 (NIH)
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Results first posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Human Immunodeficiency Virus; Acquired Immunodeficiency Syndrome; HIV Infections; Sexually Transmitted Diseases, Viral; Retroviridae Infections; Virus Diseases; Virus-HIV; RNA Virus Infections
Keywords: HIV/AIDS; Social Networks; Behavioral Economics; Incentives; PrEP; HIV Self-Testing; Fishermen; Sub Saharan Africa; Men; HIV Prevention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections; Sexually Transmitted Diseases, Viral; Retroviridae Infections; Virus Diseases; RNA Virus Infections; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Intervention Model Description: The study design is a cluster randomized controlled trial where the unit of randomization will be a clusters of men's close social network in study communities.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Promoter training, multiple self-test kits, and incentives (Experimental): Promoters in the intervention group will receive HIVST training, multiple HIVST for distribution to other men, and a small amount of remuneration (transport voucher) for themselves and to distribute to men in their networks.
  Interventions: Behavioral: Provision of multiple self-tests; Other: Small monetary incentives; Behavioral: Use of SMS/text reminders to motivate adherence to ART or PrEP
- Short training and referral for testing (No Intervention): Promoters in the control group will a short training on the basics of HIV prevention and treatment and will be encouraged to refer men in their networks for standard of care testing at the local health facilities- this may include HIV testing with a counselor or HIV self-test from the local health clinic, depending on what is available.

INTERVENTIONS:
Behavioral: Provision of multiple self-tests — Participants will be given multiple Oraquick Advance HIV-1/2 test kits for testing themselves more frequently and for men in their social networks.
  Arms: Promoter training, multiple self-test kits, and incentives
Other: Small monetary incentives — Use of small incentive voucher (~$5) to encourage linkage to confirmatory testing.
  Arms: Promoter training, multiple self-test kits, and incentives
Behavioral: Use of SMS/text reminders to motivate adherence to ART or PrEP — Messages will be motivational, will not include any identifying information and will include generic texts such as "maintain your good health", to cater for status-neutral language that can work for both HIV positive individuals taking ARVs, as well as HIV-negative individuals on PrEP who may need adherence support.
  Arms: Promoter training, multiple self-test kits, and incentives

SUMMARY:
This is a randomized controlled trial to test a combination behavioral and biomedical interventions to improve the HIV prevention and care cascades in a population of mobile men in a high priority setting (fishermen in Kenya). The intervention strategy is to recruit and train highly socially-connected men to distribute HIV self-tests and provide linkage support to men in their close social networks. The study will determine whether this social network-based approach along with small financial incentives in the form of transport vouchers can increase men's self-testing, linkage to and uptake of ART and PrEP after self-testing, virologic suppression at 6 months (for those initiating ART) and PrEP adherence (for those initiating PrEP) at 6 months. The study includes a longitudinal qualitative and mixed methods (quantitative and qualitative assessments) to identify the pathways of intervention action, and understand how the social network-based approach with support for linkage affects testing and ART and PrEP uptake and retention in men.

DETAILED DESCRIPTION:
In Aim 1, following the study pilot, community selection, and preparation the investigators will conduct a census/BMU registry verification in study communities to identify the population of men eligible for the study. The study will screen, recruit and enroll eligible men who give their informed consent to participate, then measure their close social networks identify network-central, highly-connected men ("promoters") and randomize their close social network (a cluster) to 1:1 intervention and control groups. Investigators will then conduct a baseline survey to collect socio demographic and baseline sexual behavior data among men in the close social networks. Following this baseline data collection, all promoters will be provided a training. Promoters in the intervention group will receive HIVST training, multiple HIVST for distribution to other men, and a small amount of remuneration. Promoters in the control group will receive basic HIV education and training about the study, and will be given vouchers that can be exchanged for HIV tests (standard or free HIVST kits) at nearby health facilities. Using follow-up survey data, investigators will test the hypothesis that a higher rate of HIV testing will be observed after 3 months among men in networks that receive the intervention compared to control.

In Aim 2, investigators will test whether network-central promoters can enhance linkage to ART and PrEP after HIV testing among men in their close social networks. Promoters in the Aim 1 intervention group will be asked to distribute information and transport vouchers for ART or PrEP when distributing HIV self-tests to men in their close social networks. Investigators will use clinic data to test the primary hypothesis that the intervention will result in higher rates of linkage to ART or PrEP (confirmatory testing and ART referral for positives, and PrEP screening for negatives). Investigators also will test the hypothesis that higher ART and PrEP uptake will be observed within 3 months (+ about one month) in the intervention group.

In Aim 3, investigators will measure 6 month VL and 6 month tenofovir levels using viral load testing and a novel point of care PrEP adherence assay (an antibody-based assay permitting measurement of tenofovir levels in urine) in study sites, and test the hypothesis that higher rates of virologic suppression will be observed in HIV-infected men, and PrEP adherence in un-infected men, in the intervention group. Viral load measurements will be conducted by drawing additional venous blood during routine blood draws scheduled for MOH viral load monitoring (as well as additional draws during scheduled appointments for those occurring outside of the annual VL testing standard of care window). PrEP adherence will be measured utilizing the study urine assay at 6 months. HIV treatment adherence will measured through adherence assessment during 3 and 6 routine clinic visits.

Across all aims, investigators will assess the pathways of intervention action using qualitative and mixed methods. Investigators will identify the mechanisms of action, and barriers and facilitators of the social network and incentives intervention implementation, using qualitative and mixed methods quantitative and qualitative assessments embedded in Aims 1, 2 and 3. The data collection approach will include in-depth interviews with participants in both groups, key informant interviews with network-central promoters, and focus group discussions with study participants stratified by HIV status and study group. Data will be collected at baseline and three follow-up periods corresponding to the timing of quantitative outcome measurements in Aims 1 through 3.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years or older)
* Male
* Working as a fisherman or fishing-related occupation
* Willing and able to provide informed consent for participation
* Not participating in another research study related to HIV testing, treatment and/or prevention

Exclusion Criteria:

* Younger than 18 years of age
* Female
* Included in another intervention study on HIV/AIDS
* Inadequate cognitive and/or hearing capacity to complete planned study procedures, at the discretion of the study team

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 934 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol S Camlin, MPH, PhD, Principal Investigator — University of California, San Francisco; Harsha Thirumurthy, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Impact Research Development Organization, Siaya, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] UNAIDS. 90-90-90: An ambitious treatment target to help end the AIDS epidemic. Geneva: UNAIDS;2014
- [Background] UNAIDS. THE GAP REPORT. Geneva, Switzerland 2014.
- [Background] Kwena ZA, Njuguna SW, Ssetala A, Seeley J, Nielsen L, De Bont J, Bukusi EA; Lake Victoria Consortium for Health Research (LVCHR) Team. HIV prevalence, spatial distribution and risk factors for HIV infection in the Kenyan fishing communities of Lake Victoria. PLoS One. 2019 Mar 25;14(3):e0214360. doi: 10.1371/journal.pone.0214360. eCollection 2019. PMID 30908555
- [Background] Maman D, Zeh C, Mukui I, Kirubi B, Masson S, Opolo V, Szumilin E, Riche B, Etard JF. Cascade of HIV care and population viral suppression in a high-burden region of Kenya. AIDS. 2015 Jul 31;29(12):1557-65. doi: 10.1097/QAD.0000000000000741. PMID 26244395
- [Background] NACC-NASCOP. Kenya AIDS epidemic update 2011. Nairobi, Kenya: NACC-NASCOP;2012.
- [Background] Odongo SF, Kwaro D, Mutai K. Are fisherfolk at higher risk than their neighbors: Findings from western Kenya, 2015. CROI; March 4-7, 2018; Boston, Massachusetts.
- [Background] Hoshi T, Fuji Y, Nzou SM, Tanigawa C, Kiche I, Mwau M, Mwangi AW, Karama M, Hirayama K, Goto K, Kaneko S. Spatial Distributions of HIV Infection in an Endemic Area of Western Kenya: Guiding Information for Localized HIV Control and Prevention. PLoS One. 2016 Feb 10;11(2):e0148636. doi: 10.1371/journal.pone.0148636. eCollection 2016. PMID 26862764
- [Background] Kiwanuka N, Ssetaala A, Nalutaaya A, Mpendo J, Wambuzi M, Nanvubya A, Sigirenda S, Kitandwe PK, Nielsen LE, Balyegisawa A, Kaleebu P, Nalusiba J, Sewankambo NK. High incidence of HIV-1 infection in a general population of fishing communities around Lake Victoria, Uganda. PLoS One. 2014 May 27;9(5):e94932. doi: 10.1371/journal.pone.0094932. eCollection 2014. PMID 24866840
- [Background] Asiki G, Mpendo J, Abaasa A, Agaba C, Nanvubya A, Nielsen L, Seeley J, Kaleebu P, Grosskurth H, Kamali A. HIV and syphilis prevalence and associated risk factors among fishing communities of Lake Victoria, Uganda. Sex Transm Infect. 2011 Oct;87(6):511-5. doi: 10.1136/sti.2010.046805. Epub 2011 Aug 10. PMID 21835763
- [Background] Cassels S, Camlin CS. Geographical mobility and heterogeneity of the HIV epidemic. Lancet HIV. 2016 Aug;3(8):e339-e341. doi: 10.1016/S2352-3018(16)30048-0. Epub 2016 Jul 9. No abstract available. PMID 27470023
- [Background] Kwena ZA, Bukusi EA, Ng'ayo MO, Buffardi AL, Nguti R, Richardson B, Sang NM, Holmes K. Prevalence and risk factors for sexually transmitted infections in a high-risk occupational group: the case of fishermen along Lake Victoria in Kisumu, Kenya. Int J STD AIDS. 2010 Oct;21(10):708-13. doi: 10.1258/ijsa.2010.010160. PMID 21139150
- [Background] Camlin CS, Kwena ZA, Dworkin SL. Jaboya vs. jakambi: Status, negotiation, and HIV risks among female migrants in the "sex for fish" economy in Nyanza Province, Kenya. AIDS Educ Prev. 2013 Jun;25(3):216-31. doi: 10.1521/aeap.2013.25.3.216. PMID 23631716
- [Background] Camlin CS, Kwena ZA, Dworkin SL, Cohen CR, Bukusi EA. "She mixes her business": HIV transmission and acquisition risks among female migrants in western Kenya. Soc Sci Med. 2014 Feb;102:146-56. doi: 10.1016/j.socscimed.2013.11.004. Epub 2013 Nov 15. PMID 24565152
- [Background] Fiorella KJ, Camlin CS, Salmen CR, et al. Transactional Fish-for-Sex Relationships Amid Declining Fish Access in Kenya. World Development. 2015;74:323-332.
- [Background] Kwena ZA, Camlin CS, Shisanya CA, Mwanzo I, Bukusi EA. Short-term mobility and the risk of HIV infection among married couples in the fishing communities along Lake Victoria, Kenya. PLoS One. 2013;8(1):e54523. doi: 10.1371/journal.pone.0054523. Epub 2013 Jan 15. PMID 23336005
- [Background] Camlin CS, Ssemmondo E, Chamie G, El Ayadi AM, Kwarisiima D, Sang N, Kabami J, Charlebois E, Petersen M, Clark TD, Bukusi EA, Cohen CR, R Kamya M, Havlir D; SEARCH Collaboration. Men "missing" from population-based HIV testing: insights from qualitative research. AIDS Care. 2016;28 Suppl 3(Suppl 3):67-73. doi: 10.1080/09540121.2016.1164806. PMID 27421053
- [Background] Sileo KM, Wanyenze RK, Kizito W, Reed E, Brodine SK, Chemusto H, Musoke W, Mukasa B, Kiene SM. Multi-level Determinants of Clinic Attendance and Antiretroviral Treatment Adherence Among Fishermen Living with HIV/AIDS in Communities on Lake Victoria, Uganda. AIDS Behav. 2019 Feb;23(2):406-417. doi: 10.1007/s10461-018-2207-1. PMID 29959718
- [Background] Seeley JA, Allison EH. HIV/AIDS in fishing communities: challenges to delivering antiretroviral therapy to vulnerable groups. AIDS Care. 2005 Aug;17(6):688-97. doi: 10.1080/09540120412331336698. PMID 16036255
- [Background] Johnson C, Baggaley R, Forsythe S, van Rooyen H, Ford N, Napierala Mavedzenge S, Corbett E, Natarajan P, Taegtmeyer M. Realizing the potential for HIV self-testing. AIDS Behav. 2014 Jul;18 Suppl 4:S391-5. doi: 10.1007/s10461-014-0832-x. PMID 24986599
- [Background] Napierala Mavedzenge S, Baggaley R, Corbett EL. A review of self-testing for HIV: research and policy priorities in a new era of HIV prevention. Clin Infect Dis. 2013 Jul;57(1):126-38. doi: 10.1093/cid/cit156. Epub 2013 Mar 13. PMID 23487385
- [Background] Thirumurthy H, Masters SH, Mavedzenge SN, Maman S, Omanga E, Agot K. Promoting male partner HIV testing and safer sexual decision making through secondary distribution of self-tests by HIV-negative female sex workers and women receiving antenatal and post-partum care in Kenya: a cohort study. Lancet HIV. 2016 Jun;3(6):e266-74. doi: 10.1016/S2352-3018(16)00041-2. Epub 2016 Apr 8. PMID 27240789
- [Background] Masters SH, Agot K, Obonyo B, Napierala Mavedzenge S, Maman S, Thirumurthy H. Promoting Partner Testing and Couples Testing through Secondary Distribution of HIV Self-Tests: A Randomized Clinical Trial. PLoS Med. 2016 Nov 8;13(11):e1002166. doi: 10.1371/journal.pmed.1002166. eCollection 2016 Nov. PMID 27824882
- [Background] Thirumurthy H, Masters SH, Rao S, Bronson MA, Lanham M, Omanga E, Evens E, Agot K. Effect of providing conditional economic compensation on uptake of voluntary medical male circumcision in Kenya: a randomized clinical trial. JAMA. 2014 Aug 20;312(7):703-11. doi: 10.1001/jama.2014.9087. PMID 25042290
- [Background] Chamie G, Schaffer EM, Ndyabakira A, Emperador DM, Kwarisiima D, Camlin CS, Havlir DV, Kahn JG, Kamya MR, Thirumurthy H. Comparative effectiveness of novel nonmonetary incentives to promote HIV testing. AIDS. 2018 Jul 17;32(11):1443-1451. doi: 10.1097/QAD.0000000000001833. PMID 29683850
- [Background] Sibanda EL, Tumushime M, Mufuka J, Mavedzenge SN, Gudukeya S, Bautista-Arredondo S, Hatzold K, Thirumurthy H, McCoy SI, Padian N, Copas A, Cowan FM. Effect of non-monetary incentives on uptake of couples' counselling and testing among clients attending mobile HIV services in rural Zimbabwe: a cluster-randomised trial. Lancet Glob Health. 2017 Sep;5(9):e907-e915. doi: 10.1016/S2214-109X(17)30296-6. PMID 28807189
- [Background] Gandhi M, Ameli N, Bacchetti P, Anastos K, Gange SJ, Minkoff H, Young M, Milam J, Cohen MH, Sharp GB, Huang Y, Greenblatt RM. Atazanavir concentration in hair is the strongest predictor of outcomes on antiretroviral therapy. Clin Infect Dis. 2011 May;52(10):1267-75. doi: 10.1093/cid/cir131. PMID 21507924
- [Background] Gandhi M, Bacchetti P, Rodrigues WC, Spinelli M, Koss CA, Drain PK, Baeten JM, Mugo NR, Ngure K, Benet LZ, Okochi H, Wang G, Vincent M. Development and Validation of an Immunoassay for Tenofovir in Urine as a Real-Time Metric of Antiretroviral Adherence. EClinicalMedicine. 2018 Aug-Sep;2-3:22-28. doi: 10.1016/j.eclinm.2018.08.004. Epub 2018 Aug 31. PMID 30906930
- [Background] Gandhi M, Bacchetti P, Spinelli MA, Okochi H, Baeten JM, Siriprakaisil O, Klinbuayaem V, Rodrigues WC, Wang G, Vincent M, Cressey TR, Drain PK. Brief Report: Validation of a Urine Tenofovir Immunoassay for Adherence Monitoring to PrEP and ART and Establishing the Cutoff for a Point-of-Care Test. J Acquir Immune Defic Syndr. 2019 May 1;81(1):72-77. doi: 10.1097/QAI.0000000000001971. PMID 30664078
- [Background] Spinelli MA, Glidden DV, Rodrigues WC, Wang G, Vincent M, Okochi H, Kuncze K, Mehrotra M, Defechereux P, Buchbinder SP, Grant RM, Gandhi M. Low tenofovir level in urine by a novel immunoassay is associated with seroconversion in a preexposure prophylaxis demonstration project. AIDS. 2019 Apr 1;33(5):867-872. doi: 10.1097/QAD.0000000000002135. PMID 30649051
- [Background] Lakon CM, Ennett ST, Norton EC. Mechanisms through which drug, sex partner, and friendship network characteristics relate to risky needle use among high risk youth and young adults. Soc Sci Med. 2006 Nov;63(9):2489-99. doi: 10.1016/j.socscimed.2006.06.015. Epub 2006 Jul 27. PMID 16875770
- [Background] Rudolph AE, Crawford ND, Latkin C, Fowler JH, Fuller CM. Individual and neighborhood correlates of membership in drug using networks with a higher prevalence of HIV in New York City (2006-2009). Ann Epidemiol. 2013 May;23(5):267-74. doi: 10.1016/j.annepidem.2013.02.006. Epub 2013 Mar 21. PMID 23523090
- [Background] Bohnert AS, Bradshaw CP, Latkin CA. A social network perspective on heroin and cocaine use among adults: evidence of bidirectional influences. Addiction. 2009 Jul;104(7):1210-8. doi: 10.1111/j.1360-0443.2009.02615.x. PMID 19563564
- [Background] El-Bassel N, Gilbert L, Wu E, Chang M. A social network profile and HIV risk among men on methadone: do social networks matter? J Urban Health. 2006 Jul;83(4):602-13. doi: 10.1007/s11524-006-9075-0. PMID 16755389
- [Background] Neblett RC, Davey-Rothwell M, Chander G, Latkin CA. Social network characteristics and HIV sexual risk behavior among urban African American women. J Urban Health. 2011 Feb;88(1):54-65. doi: 10.1007/s11524-010-9513-x. PMID 21234695
- [Background] King KM, Latkin CA, Davey-Rothwell MA. Love on lockdown: how social network characteristics predict separational concurrency among low income African-American women. J Urban Health. 2015 Jun;92(3):460-71. doi: 10.1007/s11524-015-9951-6. PMID 25820220
- [Background] Grieb SM, Davey-Rothwell M, Latkin CA. Social and sexual network characteristics and concurrent sexual partnerships among urban African American high-risk women with main sex partners. AIDS Behav. 2012 May;16(4):882-9. doi: 10.1007/s10461-011-0030-z. PMID 21861193
- [Background] Barrington C, Latkin C, Sweat MD, Moreno L, Ellen J, Kerrigan D. Talking the talk, walking the walk: social network norms, communication patterns, and condom use among the male partners of female sex workers in La Romana, Dominican Republic. Soc Sci Med. 2009 Jun;68(11):2037-44. doi: 10.1016/j.socscimed.2009.03.009. Epub 2009 Apr 6. PMID 19356834
- [Background] Ajilore O. Identifying peer effects using spatial analysis: the role of peers on risky sexual behavior. Rev Econ Househ. 2015 Sep;13(3):635-652. doi: 10.1007/s11150-013-9235-4. PMID 26300714
- [Background] Staveteig SW, S; Head S.K.; Bradley S; Nybo E. Demographic Patterns of HIV Testing Uptake in Sub-Saharan Africa. Calverton, Maryland, USA: ICF International;2013.
- [Background] Cornell M, Schomaker M, Garone DB, Giddy J, Hoffmann CJ, Lessells R, Maskew M, Prozesky H, Wood R, Johnson LF, Egger M, Boulle A, Myer L; International Epidemiologic Databases to Evaluate AIDS Southern Africa Collaboration. Gender differences in survival among adult patients starting antiretroviral therapy in South Africa: a multicentre cohort study. PLoS Med. 2012;9(9):e1001304. doi: 10.1371/journal.pmed.1001304. Epub 2012 Sep 4. PMID 22973181
- [Background] Ochieng-Ooko V, Ochieng D, Sidle JE, Holdsworth M, Wools-Kaloustian K, Siika AM, Yiannoutsos CT, Owiti M, Kimaiyo S, Braitstein P. Influence of gender on loss to follow-up in a large HIV treatment programme in western Kenya. Bull World Health Organ. 2010 Sep 1;88(9):681-8. doi: 10.2471/BLT.09.064329. Epub 2010 Apr 16. PMID 20865073
- [Background] Kranzer K, Lewis JJ, Ford N, Zeinecker J, Orrell C, Lawn SD, Bekker LG, Wood R. Treatment interruption in a primary care antiretroviral therapy program in South Africa: cohort analysis of trends and risk factors. J Acquir Immune Defic Syndr. 2010 Nov;55(3):e17-23. doi: 10.1097/QAI.0b013e3181f275fd. PMID 20827216
- [Background] Hawkins C, Chalamilla G, Okuma J, Spiegelman D, Hertzmark E, Aris E, Ewald T, Mugusi F, Mtasiwa D, Fawzi W. Sex differences in antiretroviral treatment outcomes among HIV-infected adults in an urban Tanzanian setting. AIDS. 2011 Jun 1;25(9):1189-97. doi: 10.1097/QAD.0b013e3283471deb. PMID 21505309
- [Background] Takarinda KC, Harries AD, Shiraishi RW, Mutasa-Apollo T, Abdul-Quader A, Mugurungi O. Gender-related differences in outcomes and attrition on antiretroviral treatment among an HIV-infected patient cohort in Zimbabwe: 2007-2010. Int J Infect Dis. 2015 Jan;30:98-105. doi: 10.1016/j.ijid.2014.11.009. Epub 2014 Nov 15. PMID 25462184
- [Background] Marson KG, Tapia K, Kohler P, McGrath CJ, John-Stewart GC, Richardson BA, Njoroge JW, Kiarie JN, Sakr SR, Chung MH. Male, mobile, and moneyed: loss to follow-up vs. transfer of care in an urban African antiretroviral treatment clinic. PLoS One. 2013 Oct 24;8(10):e78900. doi: 10.1371/journal.pone.0078900. eCollection 2013. PMID 24205345
- [Background] Penot P, Hema A, Bado G, Kabore F, Sore I, Sombie D, Traore JR, Guiard-Schmid JB, Fontanet A, Slama L, Bruno Sawadogo A, Laurent C. The vulnerability of men to virologic failure during antiretroviral therapy in a public routine clinic in Burkina Faso. J Int AIDS Soc. 2014 Jan 15;17(1):18646. doi: 10.7448/IAS.17.1.18646. eCollection 2014. PMID 24433983
- [Background] Mosha F, Muchunguzi V, Matee M, Sangeda RZ, Vercauteren J, Nsubuga P, Lyamuya E, Vandamme AM. Gender differences in HIV disease progression and treatment outcomes among HIV patients one year after starting antiretroviral treatment (ART) in Dar es Salaam, Tanzania. BMC Public Health. 2013 Jan 15;13:38. doi: 10.1186/1471-2458-13-38. PMID 23320567
- [Background] Kipp W, Alibhai A, Saunders LD, Senthilselvan A, Kaler A, Konde-Lule J, Okech-Ojony J, Rubaale T. Gender differences in antiretroviral treatment outcomes of HIV patients in rural Uganda. AIDS Care. 2010 Mar;22(3):271-8. doi: 10.1080/09540120903193625. PMID 20390506
- [Background] Boulle C, Kouanfack C, Laborde-Balen G, Boyer S, Aghokeng AF, Carrieri MP, Kaze S, Dontsop M, Mben JM, Koulla-Shiro S, Peytavin G, Spire B, Delaporte E, Laurent C; Stratall ANRS 12110ESTHER Study Group. Gender Differences in Adherence and Response to Antiretroviral Treatment in the Stratall Trial in Rural District Hospitals in Cameroon. J Acquir Immune Defic Syndr. 2015 Jul 1;69(3):355-64. doi: 10.1097/QAI.0000000000000604. PMID 26181708
- [Background] Tsai AC, Siedner MJ. The Missing Men: HIV Treatment Scale-Up and Life Expectancy in Sub-Saharan Africa. PLoS Med. 2015 Nov 24;12(11):e1001906. doi: 10.1371/journal.pmed.1001906. eCollection 2015 Nov. PMID 26599825
- [Background] Bor J, Rosen S, Chimbindi N, Haber N, Herbst K, Mutevedzi T, Tanser F, Pillay D, Barnighausen T. Mass HIV Treatment and Sex Disparities in Life Expectancy: Demographic Surveillance in Rural South Africa. PLoS Med. 2015 Nov 24;12(11):e1001905; discussion e1001905. doi: 10.1371/journal.pmed.1001905. eCollection 2015 Nov. PMID 26599699
- [Background] Vandormael A, Akullian A, Dobra A, de Oliveira T, Tanser F. Sharp decline in male HIV incidence in a rural South African population (2004-2015). CROI 2018; March 4-7, 2018; Boston, Massachusetts.
- [Background] DiCarlo AL, Mantell JE, Remien RH, Zerbe A, Morris D, Pitt B, Abrams EJ, El-Sadr WM. 'Men usually say that HIV testing is for women': gender dynamics and perceptions of HIV testing in Lesotho. Cult Health Sex. 2014;16(8):867-82. doi: 10.1080/13691058.2014.913812. Epub 2014 May 22. PMID 24854495
- [Background] May M, Boulle A, Phiri S, Messou E, Myer L, Wood R, Keiser O, Sterne JA, Dabis F, Egger M; IeDEA Southern Africa and West Africa. Prognosis of patients with HIV-1 infection starting antiretroviral therapy in sub-Saharan Africa: a collaborative analysis of scale-up programmes. Lancet. 2010 Aug 7;376(9739):449-57. doi: 10.1016/S0140-6736(10)60666-6. Epub 2010 Jul 15. PMID 20638120
- [Background] Braitstein P, Boulle A, Nash D, Brinkhof MW, Dabis F, Laurent C, Schechter M, Tuboi SH, Sprinz E, Miotti P, Hosseinipour M, May M, Egger M, Bangsberg DR, Low N; Antiretroviral Therapy in Lower Income Countries (ART-LINC) study group. Gender and the use of antiretroviral treatment in resource-constrained settings: findings from a multicenter collaboration. J Womens Health (Larchmt). 2008 Jan-Feb;17(1):47-55. doi: 10.1089/jwh.2007.0353. PMID 18240981
- [Background] Baker P, Dworkin SL, Tong S, Banks I, Shand T, Yamey G. The men's health gap: men must be included in the global health equity agenda. Bull World Health Organ. 2014 Aug 1;92(8):618-20. doi: 10.2471/BLT.13.132795. Epub 2014 Mar 6. No abstract available. PMID 25197149
- [Background] Mburu G, Ram M, Siu G, Bitira D, Skovdal M, Holland P. Intersectionality of HIV stigma and masculinity in eastern Uganda: implications for involving men in HIV programmes. BMC Public Health. 2014 Oct 11;14:1061. doi: 10.1186/1471-2458-14-1061. PMID 25304035
- [Background] Skovdal M, Campbell C, Madanhire C, Mupambireyi Z, Nyamukapa C, Gregson S. Masculinity as a barrier to men's use of HIV services in Zimbabwe. Global Health. 2011 May 15;7:13. doi: 10.1186/1744-8603-7-13. PMID 21575149
- [Background] Cornell M, McIntyre J, Myer L. Men and antiretroviral therapy in Africa: our blind spot. Trop Med Int Health. 2011 Jul;16(7):828-9. doi: 10.1111/j.1365-3156.2011.02767.x. Epub 2011 Mar 21. PMID 21418449
- [Background] Siu GE, Seeley J, Wight D. Dividuality, masculine respectability and reputation: how masculinity affects men's uptake of HIV treatment in rural eastern Uganda. Soc Sci Med. 2013 Jul;89:45-52. doi: 10.1016/j.socscimed.2013.04.025. Epub 2013 Apr 28. PMID 23726215
- [Background] Siu GE, Wight D, Seeley J. How a masculine work ethic and economic circumstances affect uptake of HIV treatment: experiences of men from an artisanal gold mining community in rural eastern Uganda. J Int AIDS Soc. 2012 Jun 14;15 Suppl 1(Suppl 1):1-9. doi: 10.7448/IAS.15.3.17368. PMID 22713356
- [Background] Camlin CS, Akullian A, Neilands TB, Getahun M, Eyul P, Maeri I, Ssali S, Geng E, Gandhi M, Cohen CR, Kamya MR, Odeny T, Bukusi EA, Charlebois ED. Population mobility associated with higher risk sexual behaviour in eastern African communities participating in a Universal Testing and Treatment trial. J Int AIDS Soc. 2018 Jul;21 Suppl 4(Suppl Suppl 4):e25115. doi: 10.1002/jia2.25115. PMID 30027668
- [Background] Camlin CS, Charlebois ED, Getahun M, Akatukwasa C, Atwine F, Itiakorit H, Bakanoma R, Maeri I, Owino L, Onyango A, Chamie G, Clark TD, Cohen CR, Kwarisiima D, Kabami J, Sang N, Kamya MR, Bukusi EA, Petersen ML, V Havlir D. Pathways for reduction of HIV-related stigma: a model derived from longitudinal qualitative research in Kenya and Uganda. J Int AIDS Soc. 2020 Dec;23(12):e25647. doi: 10.1002/jia2.25647. PMID 33283986
- [Background] Choko AT, Desmond N, Webb EL, Chavula K, Napierala-Mavedzenge S, Gaydos CA, Makombe SD, Chunda T, Squire SB, French N, Mwapasa V, Corbett EL. The uptake and accuracy of oral kits for HIV self-testing in high HIV prevalence setting: a cross-sectional feasibility study in Blantyre, Malawi. PLoS Med. 2011 Oct;8(10):e1001102. doi: 10.1371/journal.pmed.1001102. Epub 2011 Oct 4. PMID 21990966
- [Background] Lee VJ, Tan SC, Earnest A, Seong PS, Tan HH, Leo YS. User acceptability and feasibility of self-testing with HIV rapid tests. J Acquir Immune Defic Syndr. 2007 Aug 1;45(4):449-53. doi: 10.1097/QAI.0b013e318095a3f3. PMID 17554213
- [Background] Carballo-Dieguez A, Frasca T, Balan I, Ibitoye M, Dolezal C. Use of a rapid HIV home test prevents HIV exposure in a high risk sample of men who have sex with men. AIDS Behav. 2012 Oct;16(7):1753-60. doi: 10.1007/s10461-012-0274-2. PMID 22893194
- [Background] Thirumurthy H, Akello I, Murray K, et al. Acceptability and feasibility of a novel approach to promote HIV testing in sexual and social networks using HIV self-tests. . Paper presented at: International AIDS Society (IAS) conference2015; Vancouver, Canada.
- [Background] Choko AT, MacPherson P, Webb EL, Willey BA, Feasy H, Sambakunsi R, Mdolo A, Makombe SD, Desmond N, Hayes R, Maheswaran H, Corbett EL. Uptake, Accuracy, Safety, and Linkage into Care over Two Years of Promoting Annual Self-Testing for HIV in Blantyre, Malawi: A Community-Based Prospective Study. PLoS Med. 2015 Sep 8;12(9):e1001873. doi: 10.1371/journal.pmed.1001873. eCollection 2015 Sep. PMID 26348035
- [Background] Figueroa C, Johnson C, Verster A, Baggaley R. Attitudes and Acceptability on HIV Self-testing Among Key Populations: A Literature Review. AIDS Behav. 2015 Nov;19(11):1949-65. doi: 10.1007/s10461-015-1097-8. PMID 26054390
- [Background] Kalibala S, Tun W, Cherutich P, Nganga A, Oweya E, Oluoch P. Factors associated with acceptability of HIV self-testing among health care workers in Kenya. AIDS Behav. 2014 Jul;18 Suppl 4(Suppl 4):S405-14. doi: 10.1007/s10461-014-0830-z. PMID 24974123
- [Background] Kalibala S, Tun W, Muraah W. Feasibility and acceptability of HIV self testing among health care workers: results of a pilot programme in two hospitals in Kenya. XVIII International AIDS Conference; 18-23 July, 2010, 2010; Vienna, Austria 18-23 July.
- [Background] Consolidated Guidelines on HIV Testing Services: 5Cs: Consent, Confidentiality, Counselling, Correct Results and Connection 2015. Geneva: World Health Organization; 2015 Jul. Available from http://www.ncbi.nlm.nih.gov/books/NBK316021/ PMID 26378328
- [Background] Ingold H, Mwerinde O, Ross AL, Leach R, Corbett EL, Hatzold K, Johnson CC, Ncube G, Nyirenda R, Baggaley RC. The Self-Testing AfRica (STAR) Initiative: accelerating global access and scale-up of HIV self-testing. J Int AIDS Soc. 2019 Mar;22 Suppl 1(Suppl Suppl 1):e25249. doi: 10.1002/jia2.25249. PMID 30907517
- [Background] Guidelines on HIV Self-Testing and Partner Notification: Supplement to Consolidated Guidelines on HIV Testing Services. Geneva: World Health Organization; 2016 Dec. Available from http://www.ncbi.nlm.nih.gov/books/NBK401684/ PMID 27977094
- [Background] National AIDS and STD Control Programme. Guidelines for HIV Testing and Counselling in Kenya. In: Ministry of Public Health and Sanitation Kenya, ed: Nairobi: NASCOP; 2008.
- [Background] National AIDS and STI Control Programme. Guidelines for HIV Testing Services in Kenya. Nairobi: National AIDS Control Programme; 2015.
- [Background] Monge PR, Contractor NS. Theories of Communication Networks. New York: Oxford University Press; 2003.
- [Background] Valente TW. Social Networks and Health: Models, Methods, and Applications. New York: Oxford University Press; 2010.
- [Background] Newman M, Barabási AL, Watts D. The Structure and Dynamics of Networks. Princeton, NJ: Princeton University Press; 2006.
- [Background] Wasserman S, Faust K. Social network analysis: Methods and applications. Cambridge, U.K.: Cambridge University Press; 1994.
- [Background] Cross R, Parker A. The Hidden Power of Social Networks: Understanding How Work Really Gets Done in Organizations. Cambridge, MA: Harvard Business School Press; 2006.
- [Background] Sacerdote B. Peer effects with random assignment: Results for Dartmouth roommates. Q J Econ. 2001;116(2):681-704.
- [Background] Christakis NA, Fowler JH. The spread of obesity in a large social network over 32 years. N Engl J Med. 2007 Jul 26;357(4):370-9. doi: 10.1056/NEJMsa066082. Epub 2007 Jul 25. PMID 17652652
- [Background] Christakis NA, Fowler JH. Social Network Visualization in Epidemiology. Nor Epidemiol. 2009;19(1):5-16. PMID 22544996
- [Background] Valente TW. Network interventions. Science. 2012 Jul 6;337(6090):49-53. doi: 10.1126/science.1217330. PMID 22767921
- [Background] ILO. Decent Work for Domestic Workers. Paper presented at: 100th Session of the International Labour Conference (ILC)2012; Geneva.
- [Background] Latkin CA, Knowlton AR. Social Network Assessments and Interventions for Health Behavior Change: A Critical Review. Behav Med. 2015;41(3):90-7. doi: 10.1080/08964289.2015.1034645. PMID 26332926
- [Background] Shaya FT, Chirikov VV, Howard D, Foster C, Costas J, Snitker S, Frimpter J, Kucharski K. Effect of social networks intervention in type 2 diabetes: a partial randomised study. J Epidemiol Community Health. 2014 Apr;68(4):326-32. doi: 10.1136/jech-2013-203274. Epub 2013 Dec 2. PMID 24297971
- [Background] Sorkin DH, Mavandadi S, Rook KS, Biegler KA, Kilgore D, Dow E, Ngo-Metzger Q. Dyadic collaboration in shared health behavior change: the effects of a randomized trial to test a lifestyle intervention for high-risk Latinas. Health Psychol. 2014 Jun;33(6):566-75. doi: 10.1037/hea0000063. PMID 24884910
- [Background] Terzian E, Tognoni G, Bracco R, De Ruggieri E, Ficociello RA, Mezzina R, Pillo G; SIRS (Studio di Intervento sulla Rete Sociale [Social Network Intervention Study]) Collaborative Study Group. Social network intervention in patients with schizophrenia and marked social withdrawal: a randomized controlled study. Can J Psychiatry. 2013 Nov;58(11):622-31. doi: 10.1177/070674371305801108. PMID 24246433
- [Background] Yamanis TJ, Dervisevic E, Mulawa M, Conserve DF, Barrington C, Kajula LJ, Maman S. Social Network Influence on HIV Testing Among Urban Men in Tanzania. AIDS Behav. 2017 Apr;21(4):1171-1182. doi: 10.1007/s10461-016-1513-8. PMID 27506817
- [Background] Zheng WB, L.; Brown, L.; Sang, N.; Clark, T.; Charlebois, E.; Kamya, M.R.; Havlir, D.V.; Petersen, M. Local social network features predict HIV testing uptake in a rural Ugandan community. Conference on Retroviruses and Opportunistic Infections; 2016; Boston, MA.
- [Background] Zheng WS, N.; Chamie, G; Balzer, L.B.; Cohen, C.; Clark, T.D.; Charlebois, E.D.; Kamya, M.R.; Havlir, D.V.; Petersen, M. L. Social Networks and HIV Prevalence in the SEARCH Study. Conference on Retroviruses and Opportunistic Infections; 2017; Seattle, WA.
- [Background] Yamanis TJ, Fisher JC, Moody JW, Kajula LJ. Young Men's Social Network Characteristics and Associations with Sexual Partnership Concurrency in Tanzania. AIDS Behav. 2016 Jun;20(6):1244-55. doi: 10.1007/s10461-015-1152-5. PMID 26271813
- [Background] Mulawa M, Yamanis TJ, Hill LM, Balvanz P, Kajula LJ, Maman S. Evidence of social network influence on multiple HIV risk behaviors and normative beliefs among young Tanzanian men. Soc Sci Med. 2016 Mar;153:35-43. doi: 10.1016/j.socscimed.2016.02.002. Epub 2016 Feb 2. PMID 26874081
- [Background] Medley A, Kennedy C, O'Reilly K, Sweat M. Effectiveness of peer education interventions for HIV prevention in developing countries: a systematic review and meta-analysis. AIDS Educ Prev. 2009 Jun;21(3):181-206. doi: 10.1521/aeap.2009.21.3.181. PMID 19519235
- [Background] Simoni JM, Nelson KM, Franks JC, Yard SS, Lehavot K. Are peer interventions for HIV efficacious? A systematic review. AIDS Behav. 2011 Nov;15(8):1589-95. doi: 10.1007/s10461-011-9963-5. PMID 21598034
- [Background] Valente TW, Davis RL. Accelerating the diffusion of innovations using opinion leaders. Ann Am Acad Polit Ss. 1999;566:55-67.
- [Background] Kempe D, Kleinberg J, Tardos É. Maximizing the spread of influence through a social network. Theory of Computing. 2015;11(Article 4):105-147.
- [Background] Kim DA, Hwong AR, Stafford D, Hughes DA, O'Malley AJ, Fowler JH, Christakis NA. Social network targeting to maximise population behaviour change: a cluster randomised controlled trial. Lancet. 2015 Jul 11;386(9989):145-53. doi: 10.1016/S0140-6736(15)60095-2. Epub 2015 May 4. PMID 25952354
- [Background] Flodgren G, Parmelli E, Doumit G, Gattellari M, O'Brien MA, Grimshaw J, Eccles MP. Local opinion leaders: effects on professional practice and health care outcomes. Cochrane Database Syst Rev. 2011 Aug 10;(8):CD000125. doi: 10.1002/14651858.CD000125.pub4. PMID 21833939
- [Background] Baeten JM, Donnell D, Ndase P, Mugo NR, Campbell JD, Wangisi J, Tappero JW, Bukusi EA, Cohen CR, Katabira E, Ronald A, Tumwesigye E, Were E, Fife KH, Kiarie J, Farquhar C, John-Stewart G, Kakia A, Odoyo J, Mucunguzi A, Nakku-Joloba E, Twesigye R, Ngure K, Apaka C, Tamooh H, Gabona F, Mujugira A, Panteleeff D, Thomas KK, Kidoguchi L, Krows M, Revall J, Morrison S, Haugen H, Emmanuel-Ogier M, Ondrejcek L, Coombs RW, Frenkel L, Hendrix C, Bumpus NN, Bangsberg D, Haberer JE, Stevens WS, Lingappa JR, Celum C; Partners PrEP Study Team. Antiretroviral prophylaxis for HIV prevention in heterosexual men and women. N Engl J Med. 2012 Aug 2;367(5):399-410. doi: 10.1056/NEJMoa1108524. Epub 2012 Jul 11. PMID 22784037
- [Background] Van Damme L, Corneli A, Ahmed K, Agot K, Lombaard J, Kapiga S, Malahleha M, Owino F, Manongi R, Onyango J, Temu L, Monedi MC, Mak'Oketch P, Makanda M, Reblin I, Makatu SE, Saylor L, Kiernan H, Kirkendale S, Wong C, Grant R, Kashuba A, Nanda K, Mandala J, Fransen K, Deese J, Crucitti T, Mastro TD, Taylor D; FEM-PrEP Study Group. Preexposure prophylaxis for HIV infection among African women. N Engl J Med. 2012 Aug 2;367(5):411-22. doi: 10.1056/NEJMoa1202614. Epub 2012 Jul 11. PMID 22784040
- [Background] Grant RM, Lama JR, Anderson PL, McMahan V, Liu AY, Vargas L, Goicochea P, Casapia M, Guanira-Carranza JV, Ramirez-Cardich ME, Montoya-Herrera O, Fernandez T, Veloso VG, Buchbinder SP, Chariyalertsak S, Schechter M, Bekker LG, Mayer KH, Kallas EG, Amico KR, Mulligan K, Bushman LR, Hance RJ, Ganoza C, Defechereux P, Postle B, Wang F, McConnell JJ, Zheng JH, Lee J, Rooney JF, Jaffe HS, Martinez AI, Burns DN, Glidden DV; iPrEx Study Team. Preexposure chemoprophylaxis for HIV prevention in men who have sex with men. N Engl J Med. 2010 Dec 30;363(27):2587-99. doi: 10.1056/NEJMoa1011205. Epub 2010 Nov 23. PMID 21091279
- [Background] Marrazzo JM, Ramjee G, Richardson BA, Gomez K, Mgodi N, Nair G, Palanee T, Nakabiito C, van der Straten A, Noguchi L, Hendrix CW, Dai JY, Ganesh S, Mkhize B, Taljaard M, Parikh UM, Piper J, Masse B, Grossman C, Rooney J, Schwartz JL, Watts H, Marzinke MA, Hillier SL, McGowan IM, Chirenje ZM; VOICE Study Team. Tenofovir-based preexposure prophylaxis for HIV infection among African women. N Engl J Med. 2015 Feb 5;372(6):509-18. doi: 10.1056/NEJMoa1402269. PMID 25651245
- [Background] Thigpen MC, Kebaabetswe PM, Paxton LA, Smith DK, Rose CE, Segolodi TM, Henderson FL, Pathak SR, Soud FA, Chillag KL, Mutanhaurwa R, Chirwa LI, Kasonde M, Abebe D, Buliva E, Gvetadze RJ, Johnson S, Sukalac T, Thomas VT, Hart C, Johnson JA, Malotte CK, Hendrix CW, Brooks JT; TDF2 Study Group. Antiretroviral preexposure prophylaxis for heterosexual HIV transmission in Botswana. N Engl J Med. 2012 Aug 2;367(5):423-34. doi: 10.1056/NEJMoa1110711. Epub 2012 Jul 11. PMID 22784038
- [Background] Choopanya K, Martin M, Suntharasamai P, Sangkum U, Mock PA, Leethochawalit M, Chiamwongpaet S, Kitisin P, Natrujirote P, Kittimunkong S, Chuachoowong R, Gvetadze RJ, McNicholl JM, Paxton LA, Curlin ME, Hendrix CW, Vanichseni S; Bangkok Tenofovir Study Group. Antiretroviral prophylaxis for HIV infection in injecting drug users in Bangkok, Thailand (the Bangkok Tenofovir Study): a randomised, double-blind, placebo-controlled phase 3 trial. Lancet. 2013 Jun 15;381(9883):2083-90. doi: 10.1016/S0140-6736(13)61127-7. Epub 2013 Jun 13. PMID 23769234
- [Background] Corneli A, Perry B, McKenna K, Agot K, Ahmed K, Taylor J, Malamatsho F, Odhiambo J, Skhosana J, Van Damme L. Participants' Explanations for Nonadherence in the FEM-PrEP Clinical Trial. J Acquir Immune Defic Syndr. 2016 Apr 1;71(4):452-61. doi: 10.1097/QAI.0000000000000880. PMID 26536315
- [Background] van der Straten A, Stadler J, Montgomery E, Hartmann M, Magazi B, Mathebula F, Schwartz K, Laborde N, Soto-Torres L. Women's experiences with oral and vaginal pre-exposure prophylaxis: the VOICE-C qualitative study in Johannesburg, South Africa. PLoS One. 2014 Feb 21;9(2):e89118. doi: 10.1371/journal.pone.0089118. eCollection 2014. PMID 24586534
- [Background] Carroll JJ, Heffron R, Mugo N, Ngure K, Ndase P, Asiimwe S, Celum C, Baeten JM. Perceived Risk Among Human Immunodeficiency Virus Serodiscordant Couples in East Africa Taking Oral Pre-Exposure Prophylaxis. Sex Transm Dis. 2016 Aug;43(8):471-5. doi: 10.1097/OLQ.0000000000000472. PMID 27419812
- [Background] Petersen M, Balzer L, Kwarsiima D, Sang N, Chamie G, Ayieko J, Kabami J, Owaraganise A, Liegler T, Mwangwa F, Kadede K, Jain V, Plenty A, Brown L, Lavoy G, Schwab J, Black D, van der Laan M, Bukusi EA, Cohen CR, Clark TD, Charlebois E, Kamya M, Havlir D. Association of Implementation of a Universal Testing and Treatment Intervention With HIV Diagnosis, Receipt of Antiretroviral Therapy, and Viral Suppression in East Africa. JAMA. 2017 Jun 6;317(21):2196-2206. doi: 10.1001/jama.2017.5705. PMID 28586888
- [Background] Chamie G, Clark TD, Kabami J, Kadede K, Ssemmondo E, Steinfeld R, Lavoy G, Kwarisiima D, Sang N, Jain V, Thirumurthy H, Liegler T, Balzer LB, Petersen ML, Cohen CR, Bukusi EA, Kamya MR, Havlir DV, Charlebois ED. A hybrid mobile approach for population-wide HIV testing in rural east Africa: an observational study. Lancet HIV. 2016 Mar;3(3):e111-9. doi: 10.1016/S2352-3018(15)00251-9. Epub 2016 Jan 26. PMID 26939734
- [Background] Koss CA, Ayieko J, Mwangwa F, Owaraganise A, Kwarisiima D, Balzer LB, Plenty A, Sang N, Kabami J, Ruel TD, Black D, Camlin CS, Cohen CR, Bukusi EA, Clark TD, Charlebois ED, Petersen ML, Kamya MR, Havlir DV; SEARCH Collaboration. Early Adopters of Human Immunodeficiency Virus Preexposure Prophylaxis in a Population-based Combination Prevention Study in Rural Kenya and Uganda. Clin Infect Dis. 2018 Nov 28;67(12):1853-1860. doi: 10.1093/cid/ciy390. PMID 29741594
- [Background] Blumenthal J, Haubrich R. Pre-exposure prophylaxis for HIV infection: how antiretroviral pharmacology helps to monitor and improve adherence. Expert Opin Pharmacother. 2013 Sep;14(13):1777-85. doi: 10.1517/14656566.2013.812072. Epub 2013 Jun 26. PMID 23800167
- [Background] Laibson D. Golden Eggs and Hyperbolic Discounting. Quarterly Journal of Economics. 1997(112):2.
- [Background] O'Donoghue T, Rabin M. Doing it now or later. Am Econ Rev. 1999;89(1):103-124.
- [Background] Mani A, Mullainathan S, Shafir E, Zhao J. Poverty impedes cognitive function. Science. 2013 Aug 30;341(6149):976-80. doi: 10.1126/science.1238041. PMID 23990553
- [Background] Loewenstein G, Brennan T, Volpp KG. Asymmetric paternalism to improve health behaviors. JAMA. 2007 Nov 28;298(20):2415-7. doi: 10.1001/jama.298.20.2415. No abstract available. PMID 18042920
- [Background] Volpp KG, Pauly MV, Loewenstein G, Bangsberg D. P4P4P: an agenda for research on pay-for-performance for patients. Health Aff (Millwood). 2009 Jan-Feb;28(1):206-14. doi: 10.1377/hlthaff.28.1.206. PMID 19124872
- [Background] Lagarde M, Haines A, Palmer N. Conditional cash transfers for improving uptake of health interventions in low- and middle-income countries: a systematic review. JAMA. 2007 Oct 24;298(16):1900-10. doi: 10.1001/jama.298.16.1900. PMID 17954541
- [Background] Banerjee AV, Duflo E, Glennerster R, Kothari D. Improving immunisation coverage in rural India: clustered randomised controlled evaluation of immunisation campaigns with and without incentives. BMJ. 2010 May 17;340:c2220. doi: 10.1136/bmj.c2220. PMID 20478960
- [Background] Korte JE, Kisa R, Vrana-Diaz CJ, Malek AM, Buregyeya E, Matovu JKB, Kagaayi J, Musoke W, Chemusto H, Mukama SC, Ndyanabo A, Mugerwa S, Wanyenze RK. HIV Oral Self-Testing for Male Partners of Women Attending Antenatal Care in Central Uganda: Uptake of Testing and Linkage to Care in a Randomized Trial. J Acquir Immune Defic Syndr. 2020 Jul 1;84(3):271-279. doi: 10.1097/QAI.0000000000002341. PMID 32168168
- [Background] Health KMo. The State of the Health Referral System in Kenya: Results from a Baseline Study on the Functionality of the Health Referral System in Eight Counties. MEASURE Evaluation-PIMA;2013.
- [Background] Ahn C, Heo M, Zhang S. Sample Size Calculations for Clustered and Longitudinal Outcomes in Clinical Research Boca Raton, FL: CRC Press; 2015.
- [Background] Campbell MJ, Walters SJ. How to Design, Analyse and Report Cluster Randomised Trials in Medicine and Health Related Research. Chichester, UK: Wiley; 2014.
- [Derived] Sheira LA, Ayieko B, Gutin SA, Kwena ZA, Charlebois ED, Agot K, Moody J, Olugo P, Adede D, Lewis-Kulzer J, Gandhi M, Thirumurthy H, Bukusi EA, Camlin CS. Gaps in Effective HIV Pre-exposure Prophylaxis Screening and Uptake Among Fishermen in Kenya. AIDS Behav. 2025 Nov 18:10.1007/s10461-025-04950-1. doi: 10.1007/s10461-025-04950-1. Online ahead of print. PMID 41251869
- [Derived] Camlin CS, Sheira LA, Kwena ZA, Charlebois ED, Agot K, Moody J, Ayieko B, Gutin SA, Ochung A, Olugo P, Lewis-Kulzer J, Nishimura H, Gandhi M, Bukusi EA, Thirumurthy H. The effect of a social network-based intervention to promote HIV testing and linkage to HIV services among fishermen in Kenya: a cluster-randomised trial. Lancet Glob Health. 2025 Apr;13(4):e669-e678. doi: 10.1016/S2214-109X(24)00539-4. PMID 40155104
- [Derived] Sheira LA, Kwena ZA, Charlebois ED, Agot K, Ayieko B, Gandhi M, Bukusi EA, Thirumurthy H, Camlin CS. Testing a social network approach to promote HIV self-testing and linkage to care among fishermen at Lake Victoria: study protocol for the Owete cluster randomized controlled trial. Trials. 2022 Jun 6;23(1):463. doi: 10.1186/s13063-022-06409-3. PMID 35668499

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Between June 2021 and March 2022, we enumerated 1,509 fishermen in three beach communities. Among these fishermen, 934 were mapped to social networks and comprised the intent-to-treat sample. Of these, 733 men were reached and completed a baseline survey.
Units Other Than Participants: social network clusters
Period: Overall Study
Arm/Group | Promoter Training, Multiple Self-test Kits, and Incentives | Short Training and Referral for Testing
Started | 453; 77 social network clusters (Number of participants allocated to the intervention.) | 481; 79 social network clusters (Number of participants allocated to the control arm.)
Individuals | 374; 76 social network clusters (These are number of participants who completed baseline in the intervention arm.) | 359; 79 social network clusters (These are participants in the control arm for baseline.)
Completed | 353; 74 social network clusters (Number of participants who completed 3-month follow-up.) | 313; 76 social network clusters (Number of participants who completed 3-month follow-up.)
Not Completed | 100; 3 social network clusters | 168; 3 social network clusters

BASELINE CHARACTERISTICS:
Population: A total of 733 participants in 155 social network clusters.
Units Other Than Participants: Social network clusters
Groups:
- Intervention: Promoter Training, Multiple HIV Self-test Kit Distribution, and Incentive Distribution: Promoters in the intervention group will receive HIVST training, multiple HIVST for distribution to other men, and a small amount of remuneration (transport voucher) for themselves and to distribute to men in their networks.
  Provision of multiple self-tests: Participants will be given multiple Oraquick Advance HIV-1/2 test kits for testing themselves more frequently and for men in their social networks.
  Small monetary incentives: Use of small incentive voucher (~$5) to encourage linkage to confirmatory testing.
  Use of SMS/text reminders to motivate adherence to ART or PrEP: Messages will be motivational, will not include any identifying information and will include generic texts such as "maintain your good health", to cater for status-neutral language that can work for both HIV positive individuals taking ARVs, as well as HIV-negative individuals on PrEP who may need adherence support.
- Control: Promoter Training and Referral for Testing: Promoters in the control group will a short training on the basics of HIV prevention and treatment and will be encouraged to refer men in their networks for standard of care testing at the local health facilities- this may include HIV testing with a counselor or HIV self-test from the local health clinic, depending on what is available.
- Total: Total of all reporting groups
Arm/Group | Intervention: Promoter Training, Multiple HIV Self-test Kit Distribution, and Incentive Distribution | Control: Promoter Training and Referral for Testing | Total
Number analyzed (Participants) | 374 | 359 | 733
Number analyzed (Social network clusters) | 76 | 79 | 155
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 366 | 352 | 718
  >=65 years | 8 | 7 | 15
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 34.5 [28.9 to 41.2] | 37.2 [31.9 to 43.4] | 35.5 [30.1 to 42.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 374 | 359 | 733
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 374 | 359 | 733
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Kenya | 374 | 359 | 733

OUTCOME MEASURES:

1. Primary Outcome: Self-reported HIV Testing
Description: Percentage of participants who self-report HIV testing (yes/no) within the past 3 months, measured at 3-month follow-up.
Time Frame: Up to 3 months
Population: We used cluster adjusted means
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Promoter Training, Multiple Self-test Kits, and Incentives | Short Training and Referral for Testing
Number analyzed (Participants) | 353 | 313
percentage of participants | 65.6 [59.5 to 71.7] | 31.3 [25.4 to 37.2]

2. Primary Outcome: Percentage of Participants Who Linked to a Study-affiliated Clinic Within 3 Months
Description: The percentage of participants who attended a study-affiliated clinic for HIV treatment or care within 3 months of the intervention baseline
Time Frame: Up to 3 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Promoter Training, Multiple Self-test Kits, and Incentives | Short Training and Referral for Testing
Number analyzed (Participants) | 374 | 359
percentage of participants | 67.3 [61.2 to 73.5] | 15.6 [10.9 to 20.2]

3. Secondary Outcome: Linkage to PrEP
Description: Percentage of PrEP-eligible HIV-negative participants who initiate PrEP prescription (yes/no), 3-months following confirmatory testing and eligibility screening (combined)
Time Frame: Up to 3 months
Population: We used cluster adjusted means, thus the value does not yield a whole number of participants.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Intervention: Promoter Training, Multiple HIV Self-test Kit Distribution, and Incentive Distribution | Control: Promoter Training and Referral for Testing
Number analyzed (Participants) | 257 | 57
percentage | 19.7 [13.6 to 25.8] | 19.6 [9.24 to 30.1]

4. Secondary Outcome: Adherence to PrEP (% With Detectable Tenofovir in the Urine)
Description: PrEP: Percentage of PrEP-taking HIV-negative participants who are adherent to PrEP (TFV levels of >= 1500 ng/mL) at 6 months following PrEP initiation.
Time Frame: Up to 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Intervention: Promoter Training, Multiple HIV Self-test Kit Distribution, and Incentive Distribution | Control: Promoter Training and Referral for Testing
Number analyzed (Participants) | 70 | 30
percentage of participants | 18.7 | 8.3

5. Secondary Outcome: Adherence to ART
Description: ART: Percentage of HIV-positive participants who attain viral suppression (HIV RNA <400 c/mL), 6 months following ART initiation.
Time Frame: Up to 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intervention: Promoter Training, Multiple HIV Self-test Kit Distribution, and Incentive Distribution | Control: Promoter Training and Referral for Testing
Number analyzed (Participants) | 84 | 82
percentage of participants | 35.7 [25.2 to 46.3] | 40.2 [27.0 to 53.4]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected among each participant over a period of 6 months, from baseline to follow up.
Description: Same definition
Arm/Group | Promoter Training, Multiple Self-test Kits, and Incentives | Short Training and Referral for Testing
All-Cause Mortality (participants affected / at risk) | 14/374 | 0/359
Serious Adverse Events (participants affected / at risk) | 14/374 | 0/359
Other Adverse Events (participants affected / at risk) | 1/374 | 0/359
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Promoter Training, Multiple Self-test Kits, and Incentives (N=374) | Short Training and Referral for Testing (N=359)
Death (General disorders) | 14 (14) | 0 (0) — 13 deaths and 1 fracture. All were unrelated to participation in study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Promoter Training, Multiple Self-test Kits, and Incentives (N=374) | Short Training and Referral for Testing (N=359)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-11-29): https://cdn.clinicaltrials.gov/large-docs/69/NCT04772469/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/69/NCT04772469/SAP_001.pdf